CLINICAL TRIAL: NCT07176793
Title: Preventing Type 2 Diabetes Following Gestational Diabetes: Implementation Mapping for a Multilevel Breastfeeding Support Strategy
Brief Title: Pregnancy and Postpartum Breastfeeding Support for Patients With Gestational Diabetes
Status: Not yet recruiting | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 23362821; 5P30DK092924-15 (NIH); RNG211604-12 (Other Grant/Funding Number: NIDDK)
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Gestational Diabetes Mellitus (GDM); Diabetes Type 2; Breastfeeding Continuation; Breastfeeding Support
Keywords: Gestational Diabetes; Preventing Diabetes Type 2 after GDM; Breastfeeding; Focus Groups; Implementation mapping; Breastfeeding support strategy
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2; Breast Feeding

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Panel of key informants: The informant panel will include pregnant or postpartum individuals with a diagnosis of GDM. Staff at the UC Davis Health Campus including health care providers and staff who would be involved in implementing the breastfeeding support strategy and department leadership. All participants will be ≥18 years old and able to communicate in English
  Interventions: Other: Implementation mapping to develop a multilevel health system strategy for prevention of type 2 diabetes through targeted breastfeeding support for patients with gestational diabetes

INTERVENTIONS:
Other: Implementation mapping to develop a multilevel health system strategy for prevention of type 2 diabetes through targeted breastfeeding support for patients with gestational diabetes — Conduct implementation mapping to develop a multilevel health system breastfeeding support strategy for patients with GDM at UC Davis Health in Sacramento, California, a large academic medical center. The study design for this mapping process will include five steps in this 1-year proposal: (1) conduct a needs and assets assessment and identify implementers; (2) identify implementation outcomes and determinants; (3) choose mechanisms of change and design implementation strategies; (4) produce implementation protocols and materials; and prepare for the final step, (5) evaluate implementation outcomes, by selecting outcome measures for a future trial . This disciplined and systematic approach to intervention development will directly inform my future directions: a mixed methods feasibility trial to pilot the implementation strategy developed here, followed by a full-scale randomized trial to test the strategy's effectiveness in reducing diabetes risk.
  Other Names: Consolidated Framework for Implementation Research

SUMMARY:
The investigators will use implementation methods to develop better breastfeeding support for patients with gestational diabetes as a way to prevent type 2 diabetes.

DETAILED DESCRIPTION:
Gestational diabetes (GDM) is common and happens in about 8 of every 100 births. GDM can cause health problems right away and later in life. People who have GDM are 10 times more likely to get diabetes later on. Breastfeeding can help prevent diabetes. If a mother breastfeeds for 12 months or more, their chance of getting type 2 diabetes goes down by 30%. For people with GDM, not breastfeeding makes it more than twice as likely they'll get type 2 diabetes compared to those who do breastfeed. Infants also benefit-being breastfed lowers their chances of getting type 1 or type 2 diabetes later in life.

There are many barriers that people with GDM experience when breastfeeding. Compared to postpartum patients without GDM, those with GDM are 38% more likely to stop breastfeeding early. Right after birth, patients with GDM are 3.5 times less likely to be breastfeeding only (no formula) when they leave the hospital.

There are ways to help people with GDM breastfeed more, like meeting with a lactation consultant, getting help over the phone, and learning about healthy eating and exercise. But these programs aren't used much outside the hospital. Clinicians need better plans to support breastfeeding for mothers with GDM.

This study will use implementation mapping and the consolidated framework for implementation research to co-design a plan that helps mothers with GDM keep breastfeeding. The study will take place at UC Davis Health in Sacramento, California over a 1-year period.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old and able to communicate in English
* Fits into one of the following:

  1. patients with GDM who are recently pregnant and/or postpartum;
  2. health care providers (nurses, physicians, lactation consultants, etc.) who would implement the strategy
  3. executive leadership

Exclusion Criteria:

* Subjects not meeting the inclusion criteria will be considered ineligible for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Gestational Diabetes Mellitus
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Design novel implementation strategies for future mixed method trial | September 2026
  Implementation mapping data will systematically inform the design of a multilevel implementation strategy to be tested in a future pilot trial. Following guidance for rigorous early-phase studies that avoid the futility of premature, underpowered trials, this design focuses on a patient-centered, informant-engaged approach within a systematic framework; with future plans to test the implementation strategy in a feasibility trial that generates proof-of-concept evidence on a primary prevention strategy for diabetes by supporting breastfeeding for patients with GDM.

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Hoyt-Austin, DO, MAS, IBCLC, Principal Investigator — UC Davis Health

IPD SHARING:
Plan to Share IPD: Undecided